CLINICAL TRIAL: NCT02493153
Title: A Prospective Study for the Effect of Cholecystectomy to the Liver in Consideration of Hepatic Steatosis 3months After Cholecystectomy With Ultrasound
Brief Title: Hepatic Steatosis After Cholecystectomy
Acronym: HSAC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sangchul Yun (Other)
Responsible Party: Sponsor-Investigator, Sangchul Yun, M.D., Ph.D, Soonchunhyang University Hospital
Organization: Soonchunhyang University Hospital (Other)
Other Study IDs: HY-2013-N
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Hepatic Steatosis
MeSH Terms: conditions — Fatty Liver | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Liver biopsy was performed during cholecystectomy using liver wedge resection in 10 patients who had provided informed consent preoperatively. All specimens were reviewed by two pathologists with single blinded method. Sections were stained with hematoxylin and eosin (H&E) and examined at X40 magnification. Steatosis was divided into four stages using the Brunt criteria.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy — Laparoscopic cholecystectomy

SUMMARY:
The investigators are very pleased to register the study entitled "A prospective study for the effect of cholecystectomy to the liver in consideration of hepatic steatosis 3months after cholecystectomy with Ultrasound".

This study deals with prospective ultrasound study about hepatic steatosis development 3 months after cholecystectomy. This study was approved by the Institutional Review Board of the local institute. From Oct, 2013 to Jul, 2014, assessment of liver changes after cholecystectomy was carried out in 82 patients with gallbladder disease. In conclusion, the investigators thought that cholecystectomy might be considered as a risk factor for hepatic steatosis.

DETAILED DESCRIPTION:
All subjects underwent a complete medical history and physi¬cal examination. Physical examination included measurements of height and weight. Subjects with a body mass index (BMI) ≥ 30 kg/m2 were considered obese. Laboratory tests included white blood cell (WBC) count, serum albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, amylase, lipase, total cholesterol, triglycerides (TG), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), and high-sensitivity C-reactive protein (hsCRP).

In order to analyze the presence and severity of hepatic steatosis, hepatic steatosis index (HSI), US and liver biopsy was used. The hepatic steatosis index (HSI) was calculated as 8 × ALT/AST + BMI +2 (if diabetes) +2 (if female gender). All patients underwent US at the time of operation and 3 months postoperatively. All US procedures were performed by one board-certified radiologist who did not have information about the patients. Procedures were done using an iU22 apparatus (Philips Ultrasound, Bothell, WA, USA) or an EUB-7500 apparatus (Hitachi, Tokyo, Japan) equipped with a 5 MHz convex transducer. For evaluation of fatty liver, the severity of liver echogenicity was categorized. Normal echogenicity was a mild and slightly diffuse increase in hepatic echogenicity with normal visualization of diaphragm and intrahepatic vessels. Moderate echogenicity was a moderately diffuse increase in hepatic echogenicity with slightly impaired visualization of diaphragm and intrahepatic vessels. Severe echogenicity was a marked increase in hepatic echogenicity with poor or nonvisualization of the intrahepatic vessel borders, diaphragm, and posterior segment of the right hepatic lobe.

Each US image was reread by the same radiologist who was blinded to the initial reading 1 month after the initial assessment to assess intraobserver variability. Liver biopsy was performed during cholecystectomy using liver wedge resection in 10 patients who had provided informed consent preoperatively. All specimens were reviewed by two pathologists with single blinded method. Sections were stained with hematoxylin and eosin (H&E) and examined at X40 magnification. Steatosis was divided into four stages using the Brunt criteria.

ELIGIBILITY:
Inclusion Criteria:

* From Oct, 2013 to Jul, 2014, patients with a presumptive diagnosis of cholelithiasis and gallbladder polyps who was cholecystectomized

Exclusion Criteria:

* inflammatory diseases; anemia; hemochromatosis; Wilson disease; autoimmune hepa-titis; primary biliary cirrhosis; sclerosing cholangitis; biliary obstruction; alpha-1 antitrypsin deficiency; ischemic cardiac or cerebrovascular disease; impaired renal function; malignan¬cies; use of estrogens, amiodarone, steroids, tamoxifen, or lipid-lowering agents; viral hepatitis (positive serum hepatitis B surface antigen and positive serum hepatitis C antibody); iron overload (transferrin saturation ≥50%); and pregnancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From Oct, 2013 to Jul, 2014, a cohort of 82 consecutive patients with cholecystectomy was prospectively collected and followed-up.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Ultrasound finding of hepatic steatosis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dongho Choi, Principal Investigator — Hanyang University College of Medicine

REFERENCES:
- [Result] Ruhl CE, Everhart JE. Relationship of non-alcoholic fatty liver disease with cholecystectomy in the US population. Am J Gastroenterol. 2013 Jun;108(6):952-8. doi: 10.1038/ajg.2013.70. Epub 2013 Apr 2. PMID 23545713
- [Derived] Yun S, Choi D, Lee KG, Kim HJ, Kang BK, Kim H, Paik SS. Cholecystectomy Causes Ultrasound Evidence of Increased Hepatic Steatosis. World J Surg. 2016 Jun;40(6):1412-21. doi: 10.1007/s00268-015-3396-7. PMID 26796885